CLINICAL TRIAL: NCT04598737
Title: Clinical Assessment of Anterior Teeth Restored With Ultra-translucent Multilayer Zirconia Versus Lithium Disilicate Laminate Veneers (Randomized Clinical Trial)
Brief Title: Assessment of Anterior Teeth Restored With Ultra-translucent Multilayer Zirconia vs Lithium Disilicate Laminate Veneers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud abd alkarim ahmed, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: multilayer zirconia laminate
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Retention, Color Match, Marginal Adaptation and Restoration Integrity
MeSH Terms: interventions — lithia disilicate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-translucent multilayer zirconia (Experimental): Ultra-translucent multilayer zirconia laminate veneer treatment
  Interventions: Procedure: Ultra-translucent multilayer zirconia
- Lithium disilicate (Experimental): Lithium disilicate laminate veneer treatment
  Interventions: Procedure: Lithium disilicate

INTERVENTIONS:
Procedure: Ultra-translucent multilayer zirconia — Ultra-translucent multilayer zirconia laminate veneer treatment
  Arms: Ultra-translucent multilayer zirconia
Procedure: Lithium disilicate — Lithium disilicate laminate veneer treatment
  Arms: Lithium disilicate

SUMMARY:
The aim of the present study is to assess the clinical performance of multilayered translucent zirconia laminate veneers versus lithium disilicate laminate veneers in terms of modified USPHS criteria for assessment of dental restorations (retention, restoration integrity, color match and marginal adaptation)

DETAILED DESCRIPTION:
inferior mechanical properties of glass ceramics necessities the continuous development and modification for materials suitable for all clinical situations

multilayered translucent zirconia provides the advantages of high mechanical properties than all glass ceramic in addition to the improved translucency in the new generations.

Therefore, the purpose of the present study is to evaluate the clinical performance of newly introduced multilayered translucent zirconia as a monolithic laminate veneer in comparison with lithium disilicate laminate veneer to determine the clinical functional and structural integrity of the restoration

ELIGIBILITY:
Inclusion Criteria:

* sufficient sound enamel thickness
* Presence of one adjacent natural teeth that doesn't need laminate to compare shade
* age range 20 to 40 years old
* non smokers
* diastema less than 2mm
* tooth fracture not exceeding incisal one third
* normal occlusion
* vital teeth
* healthy periodontal tissues

Exclusion Criteria:

* -insufficient enamel thickness
* restoration more than 40 % of tooth surface
* parafunctional habits
* deep discoloration
* sever teeth rotation
* edge to edge or deep bite
* abnormal occlusion
* bad oral hygiene

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-10-18 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Retention | 12 months follow up period
  assessment of restoration will be done for retention on the base of of modified USPHS criteria for assessment of dental restorations

SECONDARY OUTCOMES:
Restoration integrity | 12 months follow up period
  assessment of restoration will be done for restoration integrity on the base of of modified USPHS criteria for assessment of dental restorations

OTHER OUTCOMES:
Color match | 12 months follow up period
  assessment of restoration will be done for color match on the base of of modified USPHS criteria for assessment of dental restorations
Marginal adaptation | 12 months follow up period
  assessment of restoration will be done for Marginal adaptation on the base of of modified USPHS criteria for assessment of dental restorations